CLINICAL TRIAL: NCT01243099
Title: Des Re-Endothelization for In-StEnt ResTenosis. The DESERT Study
Brief Title: Prospective Study to Assess DES Re-endothelization in BMS Restenosis and De-novo Lesions
Acronym: DESERT
Status: Completed | Type: Observational
Sponsor: S.M. Misericordia Hospital (Other)
Responsible Party: Principal Investigator, Andrea Picchi, Md. PhD, S.M. Misericordia Hospital
Other Study IDs: DSR-01
Record Dates: First submitted 2010-11-15; First posted 2010-11-18 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Stable Coronary Artery Disease; Silent Myocardial Ischemia; In-stent(BMS)Restenosis; De-novo, Atherosclerotic, Coronary Lesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- In-stent (BMS) restenosis
- De-novo coronary lesion

SUMMARY:
The hypothesis of this study is that strut coverage occurs earlier when a DES is implanted to treat a BMS restenosis compared with atherosclerotic de-novo lesion. This hypothesis is supported by two different observations: first, when a DES is implanted to treat a BMS restenosis, stent struts are deployed and drugs are eluted on a soft tissue mostly characterized by extracellular matrix with a regular surface. In this case stent malposition is less likely to occur compared to atherosclerotic lesion whose surface is often more irregular and rich in calcium. Second, patients who develop in-stent restenosis after BMS implantation are likely to show a more pronounced neointima hyperplasia and, when a DES is implanted to treat restenosis, reendothelialization is likely to occur earlier. If this hypothesis was verified, duration of dual antiplatelet therapy could be shortened after DES implantation on BMS restenosis with a clinical advantage in terms of bleeding risk. Furthermore, a higher bleeding risk is often a reason for choosing a BMS instead of a DES; thus, patients presenting with BMS restenosis are likely to have a higher bleeding risk and to benefit from a shorter period of dual antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients suitable for implantation of everolimus-eluting stents (Xcience V, Xience Prime) because of stable/unstable angina or silent myocardial ischemia due to:

* Group A: single BMS restenosis (> 50% of luminal diameter)
* Group B: single de-novo lesion (> 50% of luminal diameter)

Exclusion Criteria:

* contraindications to dual antiplatelet therapy
* acute myocardial infarction within the previous 48 hours
* significant left main coronary artery disease
* reference vessel diameter < 2.5 mm,
* hemodynamic instability
* chronic kidney disease with serum creatinine > 2 mg/dl
* pregnancy
* allergy to contrast agent, everolimus, aspirin, clopidogrel
* life expectancy < 24 months
* patients with possible low adherence to medical therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paziente affected by either stable coronary artery disease or silent myocardial ischemia
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of uncovered struts evaluated by OCT analysis at six-month follow-up. | Measured will be assessed six-month after coronary angioplasty

CONTACTS AND LOCATIONS:
Locations (1):
- Misericordia Hospital, Grosseto, Italy